CLINICAL TRIAL: NCT01414998
Title: The Effect of Non-nicotine Sensorimotor Replacement on Withdrawal and Craving: Studies With Electronic and De-nicotinised Cigarettes
Brief Title: Sensorimotor Replacement With Electronic and De-nicotinised Cigarettes
Acronym: SenRep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Dunja Przulj, Prinicipal Investigator, Queen Mary University of London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: qmul1606
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Nicotine Withdrawal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stress Ball (Active Comparator): This is the active comparator for study 1
  Interventions: Behavioral: Stress Ball vs Nicotine-free E-Cigarette
- De-nicotinised Cigarette (Experimental): This will be the experimental arm for study 2
  Interventions: Behavioral: Nicotine-free E-Cigarette vs De-nicotinised Cigarette
- Nicotine-free Electronic Cigarette (1) (Experimental): This will be the experimental arm for study 1
  Interventions: Behavioral: Stress Ball vs Nicotine-free E-Cigarette
- Nicotine-free Electronic Cigarette (2) (Active Comparator): This will be the active comparator for study 2
  Interventions: Behavioral: Nicotine-free E-Cigarette vs De-nicotinised Cigarette

INTERVENTIONS:
Behavioral: Stress Ball vs Nicotine-free E-Cigarette — In a cross over design, participants will be randomly allocated to:
  1. use a stress ball for 5 minutes during a 1 hour controlled experiment. They will also use the stress ball for one day outside of the study centre.
  2. use a nicotine-free EC for 5 minutes during a 1 hour controlled experiment. They will also use the EC ad-libitum for one day outside of the study centre.
  One week later participants will complete the other arm.
  Arms: Nicotine-free Electronic Cigarette (1); Stress Ball
Behavioral: Nicotine-free E-Cigarette vs De-nicotinised Cigarette — In a cross over design, participants will be randomly allocated to:
  1. use a nicotine-free EC for 5 minutes during a 1 hour controlled experiment. They will also use the EC ad-libitum for one day outside of the study centre.
  2. smoke 1 de-nicotinised cigarette during a 1 hour controlled experiment. They will also be given a pack to smoke ad-libitum for one day outside of the study centre.
  One week later participants will complete the other arm.
  Arms: De-nicotinised Cigarette; Nicotine-free Electronic Cigarette (2)

SUMMARY:
There are currently two sensorimotor replacement products which may be of benefit in smoking cessation: de-nicotinised cigarettes (denics) and electronic cigarettes (ECs), and the purpose of this project is to investigate whether these replacements can help to alleviate tobacco withdrawal symptoms in smokers, during a period of abstinence. This project will be separated into two studies, following the same design and procedures.

Study 1 will seek to confirm the importance of sensorimotor cues by comparing the efficacy of a nicotine-free EC in alleviating withdrawal symptoms, to a behavioural distraction tool (e.g. stress ball) which provides no smoking-related cues.

Study 2 will investigate whether sensorimotor replacements which are more proximal to smoking (i.e. Denics), will be more effective in alleviating withdrawal symptoms than a replacement which only delivers some of the conditioned sensorimotor cues (i.e. ECs).

The investigators hypothesise that the EC will be more effective at reducing withdrawal symptoms compared to the stress ball in Study 1. In Study 2, it is hypothesised that the Denic will be more effective than the EC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* Smokes at least 10 cigarettes per day
* Smokes first cigarette within 1 hour of waking

Exclusion Criteria:

* pregnant or breastfeeding
* acute psychiatric illness
* currently enrolled in other research projects
* current use of ECs or Denics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Urge to smoke at 10 minutes post product use | 10 minutes
  Urges to smoke will be measured at 10 minutes after use of products

SECONDARY OUTCOMES:
Tobacco withdrawal symptom ratings over 1 hour | 1 hour
  Change withdrawal ratings one hour after product use
Tobacco withdrawal symptom ratings over one day | 1 day
  Change in tobacco withdrawal symptom ratings over a day

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Przulj, Principal Investigator — Queen Mary University of London
Locations (1):
- Tobacco Dependence Research Unit, London, United Kingdom